CLINICAL TRIAL: NCT01373151
Title: A Phase IIB , Randomized, Multi-Center, Double-Blind, Dose-Ranging, Placebo/Active Controlled Study to Evaluate the Efficacy and Safety of BMS-945429 Subcutaneous Injection With or Without Methotrexate in Subjects With Moderate to Severe Rheumatoid Arthritis With Inadequate Response to Methotrexate.
Brief Title: Phase IIB Rheumatoid Arthritis Dose Ranging Study for BMS-945429 in Subjects Who Are Not Responding to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM133-001; 2010-023956-99 (EudraCT Number)
Record Dates: First submitted 2011-06-13; First posted 2011-06-14 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — clazakizumab; Methotrexate; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Arm 1 (Placebo Comparator): BMS-945429 Placebo/BMS-945429+Methotrexate+Adalimumab Placebo
  Interventions: Drug: BMS-945429 Placebo; Biological: BMS-945429; Drug: Methotrexate; Drug: Adalimumab Placebo
- Arm 2 (Experimental): BMS-945429 + Methotrexate + Adalimumab Placebo
  Interventions: Biological: BMS-945429; Drug: Methotrexate; Drug: Adalimumab Placebo
- Arm 3 (Experimental): BMS-945429 + Methotrexate + Adalimumab Placebo
  Interventions: Biological: BMS-945429; Drug: Methotrexate; Drug: Adalimumab Placebo
- Arm 4 (Experimental): BMS-945429 + Methotrexate + Adalimumab Placebo
  Interventions: Biological: BMS-945429; Drug: Methotrexate; Drug: Adalimumab Placebo
- Arm 5 (Experimental): BMS-945429 + Methotrexate/Methotrexate Placebo + Adalimumab Placebo
  Interventions: Biological: BMS-945429; Drug: Methotrexate Placebo; Drug: Methotrexate; Drug: Adalimumab Placebo
- Arm 6 (Experimental): BMS-945429 + Methotrexate/Methotrexate Placebo+Adalimumab Placebo
  Interventions: Biological: BMS-945429; Drug: Methotrexate Placebo; Drug: Methotrexate; Drug: Adalimumab Placebo
- Arm 7 (Active Comparator): Adalimumab + Methotrexate
  Interventions: Drug: Methotrexate; Drug: Adalimumab

INTERVENTIONS:
Drug: BMS-945429 Placebo — Injection, Subcutaneous, 0 mg, Every 4 weeks, Day 1 - Week 24 only
  Arms: Arm 1
Biological: BMS-945429 — Injection, Subcutaneous, 25 mg, Every 4 weeks, Day 1 - Week 24 only
  Arms: Arm 4
Biological: BMS-945429 — Injection, Subcutaneous, 100 mg, Every 4 weeks, 48 weeks
  Arms: Arm 3; Arm 6
Biological: BMS-945429 — Injection, Subcutaneous, 200 mg, Every 4 weeks, Week 25 - Week 48
  Arms: Arm 1; Arm 4
Biological: BMS-945429 — Injection, Subcutaneous, 200 mg, Every 4 weeks, 48 weeks
  Arms: Arm 2; Arm 5
Drug: Methotrexate — Tablets, Oral, 15 mg, Weekly, Day 1 - Week 24 only
  Arms: Arm 1
Drug: Methotrexate — Tablets, Oral, 15 mg, Weekly, 48 weeks
  Arms: Arm 2; Arm 3; Arm 4; Arm 7
Drug: Methotrexate Placebo — Tablets, Oral, 0 mg, Weekly, Day 1 - Week 24 only
  Arms: Arm 5; Arm 6
Drug: Methotrexate — Tablets, Oral, 15 mg, Weekly, Week 25 - Week 48 only
  Arms: Arm 5; Arm 6
Drug: Adalimumab Placebo — Injection, Subcutaneous, 0 mg, Every 2 weeks, 48 weeks
  Arms: Arm 1; Arm 2; Arm 3; Arm 4; Arm 5; Arm 6
Drug: Adalimumab — Injection, Subcutaneous, 40 mg, Every 2 weeks, 48 weeks
  Arms: Arm 7

SUMMARY:
The purpose of this study is to determine the effective dose of BMS-945429 in subjects with inadequate response to Methotrexate in the treatment of moderate to severe Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Inadequate response to Methotrexate
* Must have been taking Methotrexate for at least 3 months at a minimal weekly dose of at least 15 mg and stable dose for 4 weeks prior to randomization
* American College of Rheumatology (ACR) global function status class 1-3
* Minimum of 6 swollen and 6 tender joints with evidence of synovitis in at least 1 hand or wrist
* High sensitivity C-reactive protein (hsCRP) ≥ 0.8 mg/dL

Exclusion Criteria:

* Previously received or currently receiving concomitant biologic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (90):
- United States (13):
  - Sun Valley Arthritis Center, Ltd., Peoria, Arizona
  - San Diego Arthritis Medical Clinic, San Diego, California
  - New England Research Associates, Llc, Trumbull, Connecticut
  - Quincy Medical Group, Quincy, Illinois
  - Rockford Orthopedic Associates, Llc., Rockford, Illinois
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Arthritis Associates Of Mississippi, Jackson, Mississippi
  - Physician Research Collaboration, Llc, Lincoln, Nebraska
  - Box Arthritis And Rheumatology Of The Carolinas, Pllc, Charlotte, North Carolina
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Seattle Rheumatology Associates, Seattle, Washington
- Argentina (5):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Córdoba
  - Local Institution, San Juan
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Hasselt
- Brazil (5):
  - Local Institution, Goiânia, Goiás
  - Local Institution, Juiz de Fora, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo
- Canada (3):
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Centre De Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Local Institution, Prague, Czechia
- France (3):
  - Local Institution, Bordeaux
  - Local Institution, Chambray-lès-Tours
  - Local Institution, Strasbourg
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Cologne
  - Local Institution, Leipzig
  - Local Institution, Würzburg
- Hungary (4):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Gyula
  - Local Institution, Veszprém
- Italy (3):
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Reggio Emilia
- Japan (14):
  - Local Institution, Chiba, Chiba
  - Local Institution, Kitakyushu-shi, Fukuoka
  - Local Institution, Higashi-hiroshima-shi, Hiroshima
  - Local Institution, Kato-shi, Hyōgo
  - Local Institution, Miyazaki, Miyazaki
  - Local Institution, Nagano, Nagano
  - Local Institution, Nagasaki, Nagasaki
  - Local Institution, Sasebo-shi, Nagasaki
  - Local Institution, Tomigusuku-shi, Okinawa
  - Local Institution, Osaka, Osaka
  - Local Institution, Shizuoka, Shizuoka
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Shinjuku-Ku, Tokyo
  - Local Institution, Toshima-ku, Tokyo
- Mexico (6):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Morelia, Michioacan
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Culiacán, Sinaloa
  - Local Institution, San Luis Potosí City
- Local Institution, Amsterdam, Netherlands
- Poland (4):
  - Local Institution, Katowice
  - Local Institution, Krakow
  - Local Institution, Poznan
  - Local Institution, Warsaw
- Russia (6):
  - Local Institution, Kazan'
  - Local Institution, Moscow
  - Local Institution, Novosibirsk
  - Local Institution, Saint Petersburg
  - Local Institution, Yaroslavl
  - Local Institution, Yekaterinburg
- South Africa (5):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Panorama, Western Cape
  - Local Institution, Pinelands, Cape Town, Western Cape
  - Local Institution, Tygerberg, Western Cape
- South Korea (2):
  - Local Institution, Daegu
  - Local Institution, Seoul
- Spain (5):
  - Local Institution, A Coruña
  - Local Institution, Madrid
  - Local Institution, Santander
  - Local Institution, Santiago de Compostela
  - Local Institution, Seville
- Taiwan (4):
  - Local Institution, Changhua
  - Local Institution, Kaohsiung City
  - Local Institution, Taichung
  - Local Institution, Taoyuan District

REFERENCES:
- [Derived] Weinblatt ME, Mease P, Mysler E, Takeuchi T, Drescher E, Berman A, Xing J, Zilberstein M, Banerjee S, Emery P. The efficacy and safety of subcutaneous clazakizumab in patients with moderate-to-severe rheumatoid arthritis and an inadequate response to methotrexate: results from a multinational, phase IIb, randomized, double-blind, placebo/active-controlled, dose-ranging study. Arthritis Rheumatol. 2015 Oct;67(10):2591-600. doi: 10.1002/art.39249. PMID 26138593
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo+MTX: BMS-945429 (Clazakizumab)Placebo/BMS-945429+Methotrexate+Adalimumab Placebo
  BMS-945429 Placebo: Injection, Subcutaneous, 0 mg, Every 4 weeks, Day 1 - Week 24 only
  BMS-945429: Injection, Subcutaneous, 200 mg, Every 4 weeks, Week 25 - Week 48
  Methotrexate: Tablets, Oral, 15 mg, Weekly, Day 1 - Week 24 only
  Adalimumab Placebo: Injection, Subcutaneous, 0 mg, Every 2 weeks, 48 weeks
- Clazakizumab(25)+MTX: BMS-945429 + Methotrexate + Adalimumab Placebo
  BMS-945429: Injection, Subcutaneous, 200 mg, Every 4 weeks, 48 weeks
  Methotrexate: Tablets, Oral, 15 mg, Weekly, 48 weeks
  Adalimumab Placebo: Injection, Subcutaneous, 0 mg, Every 2 weeks, 48 weeks
- Clazakizumab(100): BMS-945429 + Methotrexate + Adalimumab Placebo
  BMS-945429: Injection, Subcutaneous, 100 mg, Every 4 weeks, 48 weeks
  Methotrexate: Tablets, Oral, 15 mg, Weekly, 48 weeks
  Adalimumab Placebo: Injection, Subcutaneous, 0 mg, Every 2 weeks, 48 weeks
- Clazakizumab(100)+MTX: BMS-945429 + Methotrexate + Adalimumab Placebo
  BMS-945429: Injection, Subcutaneous, 25 mg, Every 4 weeks, Day 1 - Week 24 only
  BMS-945429: Injection, Subcutaneous, 200 mg, Every 4 weeks, Week 25 - Week 48
  Methotrexate: Tablets, Oral, 15 mg, Weekly, 48 weeks
  Adalimumab Placebo: Injection, Subcutaneous, 0 mg, Every 2 weeks, 48 weeks
- Clazakizumab(200): BMS-945429 + Methotrexate/Methotrexate Placebo + Adalimumab Placebo
  BMS-945429: Injection, Subcutaneous, 200 mg, Every 4 weeks, 48 weeks
  Methotrexate Placebo: Tablets, Oral, 0 mg, Weekly, Day 1 - Week 24 only
  Methotrexate: Tablets, Oral, 15 mg, Weekly, Week 25 - Week 48 only
  Adalimumab Placebo: Injection, Subcutaneous, 0 mg, Every 2 weeks, 48 weeks
- Clazakizumab(200)+MTX: BMS-945429 + Methotrexate/Methotrexate Placebo+Adalimumab Placebo
  BMS-945429: Injection, Subcutaneous, 100 mg, Every 4 weeks, 48 weeks
  Methotrexate Placebo: Tablets, Oral, 0 mg, Weekly, Day 1 - Week 24 only
  Methotrexate: Tablets, Oral, 15 mg, Weekly, Week 25 - Week 48 only
  Adalimumab Placebo: Injection, Subcutaneous, 0 mg, Every 2 weeks, 48 weeks
- ADA+MTX: Adalimumab(ADA) + Methotrexate
  Methotrexate: Tablets, Oral, 15 mg, Weekly, 48 weeks
  Adalimumab: Injection, Subcutaneous, 40 mg, Every 2 weeks, 48 weeks
Period: Period 1
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Started | 61 | 59 | 60 | 60 | 59 | 60 | 59
Completed | 56 | 59 | 56 | 59 | 54 | 56 | 59
Not Completed | 5 | 0 | 4 | 1 | 5 | 4 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 4 | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 1 | 0 | 1 | 0
Period: Period 2
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Started | 56 | 58 | 56 | 59 | 54 | 55 | 59
Completed | 47 | 57 | 52 | 54 | 52 | 55 | 54
Not Completed | 9 | 1 | 4 | 5 | 2 | 0 | 5
Not completed — Lack of Efficacy | 9 | 0 | 0 | 1 | 2 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 3 | 3 | 0 | 0 | 1
Not completed — subject request to discontinue | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX | Total
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59 | 418
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 56 | 47 | 52 | 51 | 55 | 51 | 366
  >=65 years | 7 | 3 | 13 | 8 | 8 | 5 | 8 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.03) | 47.4 (10.97) | 55.0 (12.21) | 49.9 (13.95) | 50.0 (12.53) | 46.4 (11.91) | 52.8 (11.41) | 50.4 (12.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 46 | 52 | 53 | 49 | 49 | 48 | 343
  Male | 15 | 13 | 8 | 7 | 10 | 11 | 11 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Achieving an American College of Rheumatology (ACR) 20% Response Rate
Description: The ACR20/50/70 is a composite measure defined as both improvement of 20%, 50% or 70% in the number of tender and number of swollen joints, and a 20%, 50% or 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Time Frame: At 12 Weeks
Population: All randomized and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants | 39.3 | 76.3 | 55.0 | 73.3 | 61.0 | 60.0 | 76.3

2. Secondary Outcome: Percent of Participants With ACR 20 Response
Description: as for outcome 1
Time Frame: At 24 weeks
Population: All randomized and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants | 37.7 | 81.4 | 58.3 | 65.0 | 57.6 | 66.7 | 66.1

3. Secondary Outcome: Percent of Participants Achieving ACR 50 Response Rate
Description: as for outcome 1
Time Frame: At weeks 12 and 24
Population: All randomized and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants
  12 weeks | 21.3 | 49.2 | 26.7 | 43.3 | 28.8 | 26.7 | 30.5
  24 weeks | 16.4 | 47.5 | 36.7 | 46.7 | 33.9 | 43.3 | 47.5

4. Secondary Outcome: Percent of Participants Achieving ACR 70 Response Rate
Description: as for outcome 1
Time Frame: At weeks 12 and 24
Population: All randomized and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants
  12 weeks | 8.2 | 18.6 | 13.3 | 26.7 | 11.9 | 13.3 | 11.9
  24 weeks | 6.6 | 27.1 | 16.7 | 40.0 | 25.4 | 30.0 | 18.6

5. Secondary Outcome: Mean Change From Baseline in Disease Activity as Measured by Disease Activity Score 28 C-reactive Protein (DAS28-CRP)
Description: DAS28-CRP = Disease Activity Scores 28 based on C Reactive Protein. A DAS28-CRP below 2.6 is interpreted as remission.
Time Frame: Baseline, weeks 12 and 24
Population: All randomized and treated participants (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
score on a scale
  12 weeks: number analyzed (Participants) | 52 | 54 | 55 | 56 | 50 | 54 | 54
  12 weeks | -1.15 (0.1652) | -2.65 (0.1610) | -2.29 (0.1603) | -2.68 (0.1597) | -2.34 (0.1665) | -2.52 (0.1610) | -2.04 (0.1647)
  24 weeks: number analyzed (Participants) | 43 | 56 | 50 | 51 | 47 | 53 | 49
  24 weeks | -1.69 (0.1825) | -3.01 (0.1684) | -2.60 (0.1719) | -3.06 (0.1713) | -2.55 (0.1769) | -2.95 (0.1706) | -2.52 (0.1769)

6. Secondary Outcome: Percent of Participants With Remission by DAS28-CRP
Description: DAS28-CRP = Disease Activity Scores 28 based on C Reactive Protein. A DAS28-CRP below 2.6 is interpreted as remission.
Time Frame: At weeks 12 and 24
Population: All randomized and treated participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants
  week 12 | 1.6 | 35.6 | 21.7 | 35.0 | 25.4 | 26.7 | 20.3
  week 24 | 11.5 | 49.2 | 25.0 | 40.0 | 35.6 | 41.7 | 23.7

7. Secondary Outcome: Mean Change From Baseline in Clinical Disease Activity Index (CDAI)
Description: CDAI is a composite index for assessing disease activity. CDAI is based on the simple summation of the count of swollen joint count (SCJ) (0-28) and tender joint count (TJC) (0-28) along with patient global assessment (0-10) Scale and physician global assessment (0-10) for estimating disease activity where 10 means maximal activity. The CDAI has a range from 0 to 76.
  CDAI <= 2.8 = Remission CDAI > 2.8 and <= 10 = Low Disease Activity CDAI > 10 and <= 22 = Moderate Disease Activity CDAI > 22 = High Disease Activity
Time Frame: Baseline, weeks 12 and 24
Population: All randomized and treated participants (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
score on a scale
  week 12: number analyzed (Participants) | 54 | 58 | 55 | 56 | 52 | 55 | 57
  week 12 | -14.5 (1.727) | -22.7 (1.686) | -17.7 (1.687) | -23.1 (1.701) | -19.8 (1.738) | -21.0 (1.697) | -22.4 (1.702)
  week 24: number analyzed (Participants) | 45 | 57 | 51 | 52 | 50 | 54 | 52
  week 24 | -20.3 (1.703) | -26.1 (1.587) | -22.0 (1.613) | -26.9 (1.622) | -21.7 (1.643) | -25.6 (1.606) | -26.2 (1.631)

8. Secondary Outcome: Percent of Participants With Remission by CDAI
Description: as for outcome 7
Time Frame: At weeks 12 and 24
Population: All randomized and treated subjects
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants
  week 12 | 3.3 | 11.9 | 8.3 | 8.3 | 3.4 | 3.3 | 8.5
  week 24 | 1.6 | 15.3 | 6.7 | 21.7 | 6.8 | 20.0 | 8.5

9. Secondary Outcome: Mean Change From Baseline in Simplified Disease Activity Index (SDAI)
Description: SDAI is a composite index for assessing disease activity. CDAI is based on the simple summation of the count of swollen joint count (0-28) and tender joint count (0-28) along with patient global assessment (0-10) Scale and physician global assessment (0-10) for estimating disease activity where 10 means maximal activity and C-reactive protein (0-10). The SDAI has a range from 0 to 86.
  0.0 - 3.3 = Remission 3.4 - 11.0 = Low Activity 11.1 - 26.0 = Moderate Activity 26.1 - 86.0 = High Activity
Time Frame: Baseline, weeks 12 and 24
Population: All randomized and treated subjects (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
score on a scale
  week 12: number analyzed (Participants) | 52 | 54 | 54 | 56 | 50 | 54 | 54
  week 12 | -14.5 (1.794) | -24.9 (1.749) | -20.4 (1.745) | -25.3 (1.734) | -22.2 (1.811) | -23.3 (1.747) | -23.2 (1.785)
  week 24: number analyzed (Participants) | 43 | 56 | 50 | 51 | 47 | 53 | 49
  week 24 | -20.6 (1.812) | -28.4 (1.670) | -24.5 (1.704) | -29.1 (1.698) | -23.5 (1.755) | -27.6 (1.691) | -27.6 (1.752)

10. Secondary Outcome: Percent of Participants With Remission by SDAI
Description: as for outcome 9
Time Frame: At weeks 12 and 24
Population: All randomized and treated subjects
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants
  week 12 | 1.6 | 11.9 | 8.3 | 8.3 | 6.8 | 5.0 | 10.2
  week 24 | 4.9 | 18.6 | 6.7 | 20. | 6.8 | 23.3 | 8.5

11. Secondary Outcome: Percent of Participants With Remission Rate by Boolean Definition
Description: Boolean-based definition:
  At any time point, a patient must satisfy all of the following:
  TJC ≤1 (0-28) SJC ≤1 (0-28) CRP ≤1 mg/dl Patient Global Assessment ≤1 (on a 0-10 scale)
Time Frame: At weeks 12 and 24
Population: All randomized and treated subjects
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
percentage of participants
  week 12 | 3.3 | 8.5 | 6.7 | 10. | 1.7 | 5.0 | 5.1
  week 24 | 1.6 | 10.2 | 5.0 | 13.3 | 5.1 | 18.3 | 10.2

12. Secondary Outcome: Mean Change From Baseline in Health Assessment Questionnaire (HAQ) Disability Index
Description: Patients report the amount of difficulty they have in performing 8 categories. Each category is scored on a scale ranging from 0 (performed without any difficulty) to 3 (cannot be done at all). The HAQ-DI is then calculated by summing the scores and dividing by the number of categories answered. Total score is between 0-3.0. Increasing scores indicate worse functioning with 0 indicating no functional impairment and 3 indicating complete impairment. The HAQ-DI cannot be calculated if the subject does not have scores for at least 6 categories. A response was defined as a subject with a reduction from baseline in HAQ-DI of at least 0.22.
Time Frame: Baseline, weeks 12 and 24
Population: All randomized and treated subjects (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
score on a scale
  week 12: number analyzed (Participants) | 54 | 59 | 56 | 57 | 52 | 56 | 58
  week 12 | -0.44 (0.0827) | -0.66 (0.0801) | -0.47 (0.0807) | -0.70 (0.0811) | -0.51 (0.0834) | -0.60 (0.0807) | -0.60 (0.0819)
  week 24: number analyzed (Participants) | 44 | 58 | 51 | 53 | 50 | 56 | 53
  week 24 | -0.62 (0.0861) | -0.68 (0.0806) | -0.64 (0.0823) | -0.79 (0.0823) | -0.60 (0.0840) | -0.71 (0.0811) | -0.66 (0.0833)

13. Secondary Outcome: Mean Change From Baseline in Short Form 36 (SF-36) as Measured by Physical and Mental Components
Description: The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). To score the SF-36, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Time Frame: Baseline, weeks 12 and 24
Population: All randomized and treated subjects (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
score on a scale
  Mental component (week 12): number analyzed (Participants) | 55 | 58 | 57 | 58 | 55 | 59 | 58
  Mental component (week 12) | 5.3 (1.274) | 5.9 (1.240) | 4.5 (1.251) | 7.3 (1.244) | 4.0 (1.283) | 5.7 (1.230) | 6.4 (1.250)
  Mental component (week 24): number analyzed (Participants) | 46 | 59 | 54 | 54 | 53 | 57 | 55
  Mental component (week 24) | 6.0 (1.327) | 6.4 (1.208) | 6.6 (1.247) | 7.5 (1.247) | 5.3 (1.271) | 8.0 (1.219) | 7.1 (1.246)
  Physical component (week 12): number analyzed (Participants) | 55 | 58 | 57 | 58 | 55 | 59 | 58
  Physical component (week 12) | 4.0 (1.030) | 7.5 (0.999) | 7.3 (1.010) | 9.5 (1.002) | 6.8 (1.028) | 7.3 (0.994) | 8.4 (1.006)
  Physical component (week 24): number analyzed (Participants) | 46 | 59 | 54 | 54 | 53 | 57 | 55
  Physical component (week 24) | 6.2 (1.149) | 8.6 (1.045) | 9.4 (1.080) | 10.9 (1.076) | 7.7 (1.094) | 8.2 (1.057) | 8.2 (1.077)

14. Secondary Outcome: Mean Change From Baseline in Fatigue Severity (VAS) Score
Description: A 9-item questionnaire with questions related to how fatigue interferes with certain activities and rates its severity according to a self-report scale. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
Time Frame: Baseline, weeks 12 and 24
Population: All randomized and treated subjects (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
score on a scale
  week 12: number analyzed (Participants) | 54 | 58 | 56 | 57 | 52 | 57 | 58
  week 12 | -14.3 (3.146) | -20.8 (3.060) | -19.4 (3.077) | -27.4 (3.077) | -21.7 (3.180) | -18.6 (3.056) | -26.3 (3.080)
  week 24: number analyzed (Participants) | 45 | 57 | 51 | 54 | 50 | 56 | 53
  week 24 | -12.9 (3.306) | -23.9 (3.052) | -22.3 (3.131) | -31.3 (3.103) | -17.7 (3.184) | -23.4 (3.056) | -27.0 (3.134)

15. Secondary Outcome: Mean Change From Baseline in Work Productivity and Activity Impairment Questionnaire (WPAI) Scores
Description: The WPAI yeilds four types of scores:
  1. Absenteeism (work time missed)
  2. Presenteesism (impairment at work / reduced on-the-job effectiveness)
  3. Work productivty loss (overall work impairment / absenteeism plus presenteeism)
  4. Activity Impairment WPAI outcomes are expressed as impairment percentages with each subscale score ranging from 0-100. The subscale scores are added and averaged to produce a total WPAI score between 0-100. Higher scores indicate greater impairment and less productivity.
Time Frame: Baseline, weeks 12 and 24
Population: All randomized and treated subjects (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
score on a scale
  week 12: number analyzed (Participants) | 22 | 20 | 18 | 25 | 22 | 19 | 6
  week 12 | -9.6 (3.273) | -2.2 (3.443) | -8.7 (3.673) | -12.0 (3.081) | -13.7 (3.285) | -10.0 (3.575) | -11.7 (6.281)
  week 24: number analyzed (Participants) | 18 | 20 | 17 | 25 | 21 | 19 | 7
  week 24 | -10.7 (4.033) | -1.8 (3.893) | -17.1 (4.200) | -12.1 (3.448) | -5.9 (3.788) | -12.6 (3.938) | -4.7 (6.379)

16. Secondary Outcome: Mean Change From Baseline in Radiographic (MRI) Progression of Synovitis, Osteitis (Bone Marrow Edema), Bone Erosion and Cartilage Loss (Joint-space Narrowing)
Time Frame: Baseline and week 12
Population: All randomized and treated subjects (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: cubic millimeters
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 61 | 59 | 60 | 60 | 59 | 60 | 59
cubic millimeters
  Erosion: number analyzed (Participants) | 51 | 50 | 50 | 59 | 48 | 54 | 52
  Erosion | 1.3 (0.352) | 0.4 (0.341) | 1.1 (0.356) | 0.3 (0.334) | 1.0 (0.369) | -0.2 (0.341) | -0.5 (0.348)
  Edema: number analyzed (Participants) | 51 | 51 | 50 | 59 | 50 | 54 | 52
  Edema | 0.2 (1.009) | -6.4 (0.993) | -2.6 (1.015) | -4.7 (0.998) | -4.6 (1.036) | -5.1 (0.993) | -3.1 (1.008)
  Synovitis: number analyzed (Participants) | 51 | 51 | 50 | 59 | 50 | 54 | 52
  Synovitis | -0.5 (0.436) | -2.5 (0.427) | -1.4 (0.440) | -2.2 (0.426) | -2.9 (0.447) | -2.5 (0.427) | -2.9 (0.435)
  Narrowing: number analyzed (Participants) | 51 | 50 | 50 | 59 | 48 | 54 | 52
  Narrowing | 0.1 (0.133) | -0.1 (0.130) | 0.2 (0.135) | -0.1 (0.126) | 0.1 (0.139) | 0.0 (0.129) | -0.2 (0.132)

17. Secondary Outcome: Mean Change From Baseline in Radiographic (X-ray) Progression of Joint Damage as Measured by Modified Sharp/Van Der Heijde Total Score
Description: The Sharp-van der Heijde total score ranges from 0-528. Scores for erosion range from 0 to 5 in the hands and 0 to 10 in the feet and reflect erosion size, with 0 defined as no erosion and 3 defined as a large erosion passing the midline of the joint. If there is > 1 erosion per joint, scores can be combined to give a maximum score of 5 per joint in the hands and 10 per joint in the feet (a maximum of 5 at each side of the joint). Joint space narrowing scores vary from 0 to 4 in both the hands and feet, with 0 being normal and 4 being the absence of joint space with evident ankylosis or subluxation. Gross osteolysis and pencil-in-cup change are scored separately and, if present, are assigned the maximum score for erosion and joint space narrowing for the same affected joint. Higher scores indicate increased joint damage.
Time Frame: Baseline and week 24
Population: All randomized and treated subjects (participants with missing values at each timepoint were not included)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
Number analyzed (Participants) | 44 | 59 | 54 | 54 | 53 | 53 | 54
score on a scale | 1.8 (0.353) | 0.3 (0.320) | 0.0 (0.327) | 0.1 (0.324) | 0.1 (0.330) | 0.1 (0.336) | 0.1 (0.333)

ADVERSE EVENTS:
Time Frame: Up to 48 weeks per participant
Arm/Group | Placebo+MTX | Clazakizumab(25)+MTX | Clazakizumab(100) | Clazakizumab(100)+MTX | Clazakizumab(200) | Clazakizumab(200)+MTX | ADA+MTX
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/60 | 0/60 | 0/59 | 0/60 | 0/59
Serious Adverse Events (participants affected / at risk) | 2/61 | 5/59 | 5/60 | 5/60 | 8/59 | 5/60 | 3/59
Other Adverse Events (participants affected / at risk) | 24/61 | 43/59 | 43/60 | 51/60 | 43/59 | 50/60 | 35/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+MTX (N=61) | Clazakizumab(25)+MTX (N=59) | Clazakizumab(100) (N=60) | Clazakizumab(100)+MTX (N=60) | Clazakizumab(200) (N=59) | Clazakizumab(200)+MTX (N=60) | ADA+MTX (N=59)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective tenosynovitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Traumatic haematoma (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+MTX (N=61) | Clazakizumab(25)+MTX (N=59) | Clazakizumab(100) (N=60) | Clazakizumab(100)+MTX (N=60) | Clazakizumab(200) (N=59) | Clazakizumab(200)+MTX (N=60) | ADA+MTX (N=59)
Injection site reaction (General disorders) | 0 | 8 | 9 | 11 | 14 | 9 | 1
Ejection site erythema (General disorders) | 0 | 2 | 8 | 15 | 10 | 9 | 2
Injection site rash (General disorders) | 0 | 1 | 8 | 8 | 2 | 8 | 0
Injection site dermatitis (General disorders) | 0 | 4 | 3 | 4 | 4 | 7 | 0
Asthenia (General disorders) | 2 | 1 | 0 | 0 | 1 | 3 | 1
Injection site hypersensitivity (General disorders) | 0 | 0 | 3 | 2 | 2 | 1 | 0
Injection site papule (General disorders) | 0 | 1 | 2 | 0 | 1 | 3 | 0
Injection site pruritis (General disorders) | 0 | 1 | 0 | 4 | 0 | 1 | 0
Injection site macule (General disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3
Nasopharyngitis (Infections and infestations) | 4 | 2 | 3 | 4 | 3 | 7 | 2
Upper respiraory tract infection (Infections and infestations) | 7 | 5 | 1 | 3 | 7 | 1 | 0
Pharyngitis (Infections and infestations) | 5 | 2 | 3 | 3 | 3 | 3 | 3
Urinary tract infection (Infections and infestations) | 4 | 5 | 1 | 2 | 2 | 5 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 2 | 0 | 2 | 2 | 3
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 1 | 3 | 0 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 7 | 7 | 5 | 5 | 9 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 7 | 4 | 2 | 2 | 4 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 1 | 1 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 2
Alanine aminotransferase increased (Investigations) | 2 | 11 | 2 | 13 | 1 | 18 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 8 | 0 | 14 | 0 | 12 | 2
Gamma-glutamyltransferease increased (Investigations) | 1 | 0 | 2 | 4 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 3 | 2 | 3 | 6
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0 | 1 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 4 | 2 | 4 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 2 | 4 | 3 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 4 | 6 | 2 | 2
Headache (Nervous system disorders) | 5 | 2 | 0 | 0 | 1 | 2 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 1 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 3 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No